CLINICAL TRIAL: NCT03712579
Title: Impact of High-fat Meals Varying in Fatty Acid Composition on Adipose and Systemic Metabolic-inflammatory Responses: a Randomized Controlled Postprandial Study
Brief Title: Impact of High-fat Meals Varying in Fatty Acid Composition on Adipose and Systemic Metabolic-inflammatory Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Oonagh Markey, Vice-Chancellor's Research Fellow, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R18-P124
Record Dates: First submitted 2018-06-06; First posted 2018-10-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Inflammation; Obesity; Inflammatory Response; Cardiovascular Diseases; Overweight
MeSH Terms: conditions — Inflammation; Obesity; Cardiovascular Diseases; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFA-Rich Meal (Experimental): Participants will consume a SFA-rich test meal (75g test fat) and sequential blood and white adipose tissue samples will be collected
  Interventions: Dietary Supplement: SFA-Rich Meal
- MUFA-Rich Meal (Experimental): Participants will consume a MUFA-rich test meal (75g test fat) and sequential blood and white adipose tissue samples will be collected
  Interventions: Dietary Supplement: MUFA-Rich Meal

INTERVENTIONS:
Dietary Supplement: SFA-Rich Meal — Saturated fatty acid-rich test meal, containing 75g test fat
  Arms: SFA-Rich Meal
Dietary Supplement: MUFA-Rich Meal — Monounsaturated fatty acid-rich test meal, containing 75g test fat
  Arms: MUFA-Rich Meal

SUMMARY:
Cardiometabolic disorders are a leading cause of death worldwide. Replacing saturated fatty acids (SFA) with unsaturated fatty acids is recommended as a way of lowering cardiometabolic disease risk.

Consuming a diet rich in SFA may lead to a greater metabolic-inflammatory response in white adipose tissue during the fasting state, when compared to eating a diet rich in monounsaturated fatty acids (MUFA). Since individuals spend most of the day in the fed (or postprandial) state, it is important to see how different types of dietary fatty acids affect postprandial white adipose tissue and systemic metabolic-inflammatory responses.

This study will investigate the effect of a SFA-rich meal on markers of white adipose tissue and systemic metabolic-inflammation, compared to a MUFA-rich meal in overweight adults. In a randomised, single blind controlled, cross-over manner participants will consume either a SFA- or MUFA-rich meal and sequential blood and white adipose tissue samples will be collected before and until 6 hours postprandially.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years
* BMI = 25-40 kg/m2
* Male or Female
* Waist circumference >94 cm (men) and >80cm (women)*
* Physically active (> 3 x 30 min moderate intensity exercise per week)
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* No cardiometabolic (e.g. heart disease, high blood pressure, type 2 diabetes) or inflammatory illness

  * NOTE: If waist circumference falls below 94 cm for men or 80cm for women but BMI is >25 kg/m2 volunteers may still be recruited at the PI's discretion.

Exclusion Criteria:

* Smoker
* Previous diagnosis of anaemia
* Women who are pregnant or lactating
* Taking medication known to interfere with study outcomes (e.g. treatment for hyperlidaemia, hypertension, inflammation or hypercoagulation) or prescribed antibiotics within the last 3 months
* Taking nutritional supplements known to interfere with study outcomes (e.g. fish oil or evening primrose oil)
* Unstable weight history (>3 kg loss or gain in the previous 3 months)
* An allergy to lidocaine
* Those with known or suspected food intolerances, allergies or hypersensitivity to any components of the meal (e.g. lactose/wheat intolerance)
* Alcohol consumption >28 units per week for a man or >21 units per week for a woman
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention or metabolic study
* Parallel participation in another intervention study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Protein expression (content and phosphorylation) of key markers of metabolic inflammation in white adipose tissue (for example assessment of NFKB/IKBa total protein and phosphorylation by western blot analysis) | White adipose tissue samples will be collected at -0.5 (fasted), 1, 4 and 6 hours postprandially
  This will be assessed following the collection of white adipose tissue samples across the postprandial period

SECONDARY OUTCOMES:
Systemic Markers of Inflammation (for example TNFa and IL-6 concentrations, determined using an ELISA) | Blood samples will be collected at -0.5 (fasted) until 6 hours postprandially
  This will be assessed following the collection of blood samples
Gene expression of key markers of metabolic inflammation in white adipose tissue | White adipose tissue samples will be collected at -0.5 (fasted), 1, 4 and 6 hours postprandially
  This will be assessed following the collection of white adipose tissue samples
Characterisation of immune cell populations (monocyte subsets) from peripheral blood mononuclear cells (measured using flow cytometry analysis) | Blood samples will be collected at -0.5 (fasted) and 4 hours postprandially
  Assessed following the collection of blood samples
Serum Markers of Insulin Resistance | Blood samples will be collected at -0.5 (fasted) until 6 hours postprandially
  Assessed following the collection of blood samples
Serum Lipid Profile (primarily triacylglycerol and non-esterified fatty acid concentrations, measured using a spectrophotometric assay) | Blood samples will be collected at -0.5 (fasted) until 6 hours postprandially
  Assessed following the collection of blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Oonagh Markey, BSc, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom